CLINICAL TRIAL: NCT03121781
Title: Effect of Nasal Continuous Positive Airway Pressure (nCPAP) With RAM Cannula Versus Standard Binasal Prongs on Diaphragm Electrical Activity in Very Low Birth Weight (VLBW) Preterm Infants
Brief Title: Diaphragm Electrical Activity of Preterm Infants on nCPAP With Binasal Prongs Versus RAM Cannula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAM cannula study
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2017-04

CONDITIONS: Preterm Infants; Respiratory Distress Syndrome; CPAP; RAM Cannula; Diaphragm Electrical Activity
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Randomization will be done by sealed envelopes, ready for use once consent is obtained.Each envelope will contain a card with the assigned treatment group: protocol 1 or protocol 2.
  Protocol 1: we start the study on CPAP with binasal prongs. Edi will be recorded while the infant is on nasal CPAP with the binasal prongs, with a PEEP of 5-8 cm H2O, for 2 hours. Then, the infant will be switched the interface to the RAM cannula, with a PEEP 2 cmH2O higher, during 2 hours.
  Protocol 2: we start the study on CPAP with RAM cannula. Edi will be recorded while the infant is on nasal CPAP with the RAM cannula with a PEEP 2 cmH20 higher than the levels the infant was receiving before starting the study protocol, for 2 hours. Then, the infant will be switched the interface to the binasal prongs with a PEEP between 5-8 cmH2O, during 2 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP with binasal prongs (Active Comparator): Edi will be recorded while the infant is on nasal CPAP with the binasal prongs, with a PEEP of 5-8 cm H2O, for 2 hours. Then, the infant will be switched the interface to the RAM cannula, with a PEEP 2 cmH2O higher, during 2 hours.
  Interventions: Other: respiratory support- interface
- CPAP with RAM cannula (Active Comparator): Edi will be recorded while the infant is on nasal CPAP with the RAM cannula with a PEEP 2 cmH20 higher than the levels the infant was receiving before starting the study protocol, for 2 hours. Then, the infant will be switched the interface to the binasal prongs with a PEEP between 5-8 cmH2O, during 2 hours.
  Interventions: Other: respiratory support- interface

INTERVENTIONS:
Other: respiratory support- interface — change interface to RAM cannula
  Arms: CPAP with binasal prongs
Other: respiratory support- interface — change interface to binasal prongs
  Arms: CPAP with RAM cannula

SUMMARY:
Preterm babies have immature lungs and frequent pauses in their breathing which often necessitates breathing support. Nasal Continuous Positive Airway Pressure (nCPAP) is one of the most commonly used tools, but the standard interfaces (prongs or mask) may cause nasal-septal injury and discomfort.

The RAM cannula is another interface that consists in soft and curved prongs to avoid this nasal injury, but as the seal is not 100%, suboptimal delivery of airway distending pressure could result if they are used to deliver CPAP, as compared to standard interfaces.

The investigators plan to study very low birth weight preterm babies who are generally well but require some support with their breathing. By inserting a special feeding tube with sensors into the stomach, the investigators can measure the electrical activity of the diaphragm (EAdi), which is an important muscle for breathing. By analyzing EAdi in babies receiving nCPAP either with prongs or ram cannula, the investigators will be able to measure and compare how each method of support affects a baby's breathing. This important study will help us determine the most appropriate breathing support for preterm babies.

DETAILED DESCRIPTION:
Continuous Positive Airway Pressure is one of the most researched and accepted methods of delivering NIV to term and preterm infants. Different interfaces have been used, most frequently binasal prongs or mask. The RAM cannula is a relatively new interface for delivering CPAP in preterm infants, specially to avoid nasal injury and discomfort. However, there are few studies in artificial models with different results in term of the percentage of pressure that is really delivered when we use the RAM cannula. The objective of this study is to to investigate in VLBW preterm infants who require respiratory support by nasal CPAP, whether or not using the RAM cannula as the interface will allow to provide the level of respiratory support equivalent to that with the traditional binasal prongs, measured by diaphragm electrical activity (Edi). The investigators hypothesize that in VLBW preterm infants with respiratory distress syndrome (RDS), the use of CPAP with RAM cannula as the interface may provide lower PEEP (positive end expiratory pressure) than set and increased resistance to gas flow, leading to increased respiratory effort for the patient as reflected by an increase in Edi.

This study will help Neonatologist determine if the amount of support provided with the RAM cannula as interface is equivalent to the support we achieve with the standard interfaces, to select the patients that could benefit from using this interface. The investigators will be able to utilize this information to decide on the most appropriate respiratory support modality for preterm patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable preterm infants (defined as: cardiovascular stability with normal blood pressure and heart rate for GA and no recent increase in apneic episodes or spells and confirmed by the attending neonatologist) with birth weights less than 1500 gr and/or gestational age bellow 32 weeks, admitted to the NICU at Sunnybrook Health Sciences Centre on nasal continuous positive airway pressure of 5 to 8 cmH20 support, for at least 48 h and requiring less than 35% of oxygen.

Exclusion Criteria:

* Infants with congenital anomalies of the gastrointestinal tract, phrenic nerve damage, diaphragmatic paralysis, esophageal perforation; infants with congenital or acquired neurological deficit (including significant intraventricular hemorrhage greater than Grade II), neonatal seizure; infants with significant congenital heart disease (including symptomatic PDA); infant with congenital anomalies of the diaphragm; infant with congenital anomalies of the respiratory tracts (e.g. Congenital Cystic Adenomatoid Malformation (CCAM)) infants requiring ongoing treatment for sepsis, necrotizing enterocolitis (NEC), antibiotics for lung infections, narcotic analgesics, or gastric motility agents will be excluded. Infants on nasal CPAP and requiring more than 35% oxygen will be excluded from the study. Infants with significant gastric residuals and vomiting, infants with facial anomalies, infants with pneumothorax or pneumomediastinum, and infants in the immediate postoperative period will be excluded. Infants with nasal excoriations will be excluded from the study as they may be electively placed on the RAM cannula to prevent further nasal trauma.

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in Edi min between CPAP with binasal prongs versus with the RAM cannula | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP with binasal prongs and RAM cannula)

SECONDARY OUTCOMES:
Difference in neural respiratory rate | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP with binasal prongs and RAM cannula).
Difference in neural inspiratory time | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP with binasal prongs and RAM cannula).
Difference in Edi peak | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP with binasal prongs and RAM cannula).
Difference in transcutaneous pCO2 | 4 hours
  Measured difference in transcutaneous pCO2 between the 2 different respiratory support modes(nCPAP with binasal prongs and RAM cannula).
Difference in number of apnea episodes | 4 hours
  Difference in number of apnea episodes between the 2 different respiratory support modes (nCPAP with binasal prongs and RAM cannula).
Needs of oxygen | 4 hours
  Needs of O2 measured by FiO2 on the 2 different respiratory support modes (nCPAP with binasal prongs and RAM cannula).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunn, MD, Principal Investigator — Staff Neonatologist - NICU
Locations (1):
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No